CLINICAL TRIAL: NCT04978428
Title: An Open-Label Trial of Epidiolex in the Treatment of Obsessive Compulsive Disorder and Related Disorders: Proof of Concept Study
Brief Title: Epidiolex in Obsessive Compulsive Disorder and Related Disorders
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB21-1147
Record Dates: First submitted 2021-07-20; First posted 2021-07-27 (Actual); Last update posted 2025-05-04 (Actual); Status verified 2025-05

CONDITIONS: Obsessive-Compulsive Disorder; Trichotillomania (Hair-Pulling Disorder); Tourette Syndrome; Hoarding Disorder
Keywords: Obsessive Compulsive Disorder; CBD; Hoarding; Tourettes; Trichotillomania; Skin Picking Disorder; Body focused repetitive behaviors
MeSH Terms: conditions — Obsessive-Compulsive Disorder; Trichotillomania; Tourette Syndrome; Hoarding Disorder; Hoarding; Excoriation Disorder | interventions — Cannabidiol

STUDY DESIGN:
Intervention Model Description: Open-Label treatment study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Epidiolex (Experimental): Epidiolex (2.5 mg/kg twice daily for one week) followed by Epidiolex (5mg/kg twice daily for two weeks)
  Interventions: Drug: Cannabidiol

INTERVENTIONS:
Drug: Cannabidiol — Epidiolex oral solution (2.5 mg/kg and 5 mg/kg)
  Other Names: Epidiolex

SUMMARY:
The primary objective of the proposed study is to evaluate the safety and efficacy of Epidiolex (cannabidiol) in adults with obsessive compulsive and related disorders (OCRDs). Subjects will be treated in an open-label fashion with Epidiolex for two weeks.

DETAILED DESCRIPTION:
The primary objective of the proposed study is to evaluate the safety and efficacy of Epidiolex (cannabidiol) in adults with obsessive compulsive and related disorders (OCRDs). OCRDs include obsessive compulsive disorder (OCD), trichotillomania, skin picking, tourettes disorder, and hoarding disorders. These disorders appear linked in terms of phenomenology and possibly biology. Fifteen subjects with OCRDs will be treated in an open-label fashion with Epidiolex (2.5 mg/kg twice daily for one week followed by 5mg/kg twice daily) for two total weeks of active treatment. The hypothesis to be tested is that Epidiolex will result in reduction in symptoms of OCRDs (improvement in symptoms will be indicated by lower scores on established outcome measures of OCRDs symptoms that have been used in prior studies).

ELIGIBILITY:
Inclusion Criteria:

* Men and women age 18-65
* Primary diagnosis of OCD, Hoarding Disorder, Skin Picking Disorder, Trichotillomania, or Tourette Syndrome
* YBOCS score of at least 18 at baseline
* Ability to understand and sign the consent form.

Exclusion Criteria:

* Unstable medical illness based on history or clinically significant abnormalities on baseline physical examination or labs
* Current pregnancy or lactation, or inadequate contraception in women of childbearing potential
* Subjects considered an immediate suicide risk based on the Columbia Suicide Severity Rating Scale (C-SSRS)
* Past 12-month DSM-5 psychiatric disorder other than OCD
* Illegal substance use based on urine toxicology screening
* Initiation of psychological interventions within 3 months of screening
* Use of any other psychotropic medication
* Previous treatment with Epidiolex
* Cognitive impairment that interferes with the capacity to understand and self-administer medication or provide written informed consent

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2022-04-14 (Actual); Primary Completion 2025-11 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Yale Brown Obsessive Compulsive Scale (YBOCS) | Baseline to Week 2
  The primary outcome measure will be the change from baseline using the Yale Brown Obsessive Compulsive Scale (YBOCS). The YBOCS is a 10-item scale that assesses OCD symptoms during the last seven days. The first five items comprise the urge/thought subscale and items 6-10 comprise the behavior subscale.
NIMH Symptom Severity Scale (for TTM or Skin Picking) | Baseline to Week 2
  The primary efficacy measure will be the change in hair pulling or skin picking frequency and urges to pull hair or pick skin for the past week as indicated by change in total score. The entire study lasts 10 weeks. Every two weeks subjects will take the NIMH-TSS. The change in scores from baseline to after 10 weeks will be assessed. The scale itself assesses severity of trichotillomania symptoms. The NIMH-TSS score ranges from 0 to 20, with 0 being no symptoms and 20 being the most severe.
The Hoarding Rating Scale (HRS) | Baseline to Week 2
  The Hoarding Rating Scale is a brief, clinician rated 5-item scale This tool includes 5 questions about clutter, difficulty discarding, excessive acquisition, and the resulting distress and impairment caused by hoarding. Initial studies suggest that a score of 14 or higher on the HRS indicates a probable hoarding problem/Hoarding Disorder diagnosis.
Yale Global Tic Severity Scale (YGTSS) | Baseline to Week 2
  The Yale Global Tic Severity Scale is a semi-structured clinical interview and currently the gold standard for assessing the severity of tics in children and adults. The YGTSS enables evaluations of number, frequency, intensity, complexity, and interference of motor and phonic tics, covering the past week. Each domain is scored on a 6-point scale (range 0-5) with a separate rating for "overall impairment" regarding the subject's daily life and activities (4). Five sum scores can be created: the total motor tic score (range 0-25), the total phonic tic score (range 0-25), the total tic score (TTS; sum of the total motor tic score plus the total phonic tic score), the overall impairment rating (one item; range 0-50), and the global severity score (GSS; sum of the TTS plus the overall impairment rating, range 0-100). Higher scores reflect worse severity and worse impairment.

SECONDARY OUTCOMES:
Clinical Global Impressions- Improvement Scale (CGI-I) | Baseline to Week 2
  The entire study for the subject will last 8 weeks. Every week the subject will complete the CGI. The change in scores from baseline to after 8 weeks will be assessed. The scale itself assesses overall disorder severity on a scale from 1 to 7 with 1 being "not at all" and 7 being "among the most severe cases"
Hamilton Depression Rating Scale (HAM-D) | Baseline to Week 2
  A clinician-administered assessment of depression that will be assessed at all study visits. Higher total scores indicate higher levels of depression, while a score of 0 would indicate no depressive symptoms.
Hamilton Anxiety Rating Scale (HAM-A) | Baseline to Week 2
  A clinician-administered assessment of anxiety that will be assessed at all study visits. Changes in scores from baseline to final visit will be assessed. Higher scores indicate higher levels of anxiety, with 0 being no symptoms of anxiety.
Sheehan Disability Scale (SDS) | Baseline to Week 2
  Subjects will complete the SDS at all visits. The change in scores from baseline to study completion will be assessed. The scale itself assesses the level of disability from target disorder with higher scores indicating a more debilitating disorder.
Quality of Life Inventory (QOLI) | Baseline to Week 2
  A self-report assessment of patient perceived quality of life that will be assessed at baseline and week 8. Higher scores indicate a higher quality of life, whereas lower scores indicate a lower quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Jon E Grant, MD, JD, MPH, Principal Investigator — University of Chicago
Locations (1):
- University of Chicago, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Blanco C, Olfson M, Stein DJ, Simpson HB, Gameroff MJ, Narrow WH. Treatment of obsessive-compulsive disorder by U.S. psychiatrists. J Clin Psychiatry. 2006 Jun;67(6):946-51. doi: 10.4088/jcp.v67n0611. PMID 16848654
- [Background] Bloch MH, Landeros-Weisenberger A, Kelmendi B, Coric V, Bracken MB, Leckman JF. A systematic review: antipsychotic augmentation with treatment refractory obsessive-compulsive disorder. Mol Psychiatry. 2006 Jul;11(7):622-32. doi: 10.1038/sj.mp.4001823. Epub 2006 Apr 4. PMID 16585942
- [Background] Frisch MB, Cornell J, Villaneuva M (1993). Clinical validation of the Quality of Life Inventory: a measure of life satisfaction for use in treatment planning and outcome assessment. Psychol Assess. 4:92-101.
- [Background] Grant JE. Clinical practice: Obsessive-compulsive disorder. N Engl J Med. 2014 Aug 14;371(7):646-53. doi: 10.1056/NEJMcp1402176. PMID 25119610
- [Background] HAMILTON M. A rating scale for depression. J Neurol Neurosurg Psychiatry. 1960 Feb;23(1):56-62. doi: 10.1136/jnnp.23.1.56. No abstract available. PMID 14399272
- [Background] HAMILTON M. The assessment of anxiety states by rating. Br J Med Psychol. 1959;32(1):50-5. doi: 10.1111/j.2044-8341.1959.tb00467.x. No abstract available. PMID 13638508
- [Background] Ravizza L, Barzega G, Bellino S, Bogetto F, Maina G. Predictors of drug treatment response in obsessive-compulsive disorder. J Clin Psychiatry. 1995 Aug;56(8):368-73. PMID 7635854
- [Background] Sheehan DV (1983). The Anxiety Disease. New York: Scribner's.
- [Background] Sheehan DV, Lecrubier Y, Sheehan KH, Amorim P, Janavs J, Weiller E, Hergueta T, Baker R, Dunbar GC. The Mini-International Neuropsychiatric Interview (M.I.N.I.): the development and validation of a structured diagnostic psychiatric interview for DSM-IV and ICD-10. J Clin Psychiatry. 1998;59 Suppl 20:22-33;quiz 34-57. PMID 9881538